CLINICAL TRIAL: NCT07131072
Title: A Prospective Study- Assessment of Diaphragmatic Role in Dyspneic Patients With Different Types of Interstitial Lung Disease
Brief Title: Assessment of Diaphragmatic Mobility in Dyspneic Patients With Different Types of Interstitial Lung Diseases
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, hieba gamal ezz-elragal awad, Assistant professor, Ain Shams University
Other Study IDs: FMASU R13/2021
Record Dates: First submitted 2025-08-06; First posted 2025-08-20 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Diaphragm Issues

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- collagen related interstitial lung disease
  Interventions: Other: daiphragm mobility by ultrsound; Other: spirometry ,DLCo
- idiopathic type (IPF)
  Interventions: Other: daiphragm mobility by ultrsound; Other: spirometry ,DLCo
- OTHERS(occupational,sarcoid,...)
  Interventions: Other: daiphragm mobility by ultrsound; Other: spirometry ,DLCo

INTERVENTIONS:
Other: daiphragm mobility by ultrsound — fibrosis score, alveolitis score by CT Chest
  Other Names: warricks score
Other: spirometry ,DLCo — FEV1, FVC, FEV1/FVC, DLCo

SUMMARY:
dyspnea and impaired exercise capacity in IPF patients can be related, at least in part, to respiratory muscle dysfunction, in particular to diaphragm functionality. Both B-mode and M-mode ultrasound techniques have been employed to assess diaphragm excursion, which measures the distance that the diaphragm is able to move during the respiratory cycle.

recent study using lung ultrasound in assessment of diaphragmatic mobility in IPF patients and found that Diaphragmatic mobility is lower in IPF patients than in healthy controls, especially during deep inspiration. The correlation between reduced FVC and diaphragmatic excursion values in IPF patients can be of interest, since it could represent an index of functional respiratory affection performed by chest ultrasound

DETAILED DESCRIPTION:
Interstitial lung diseases are known to be associated with limitations in daily activities and impaired quality of life. One of the most troublesome burdens for ILD patients is dyspnea during exercise, which extends to the resting state as the disease advances. The causes of dyspnea are suggested to be a progressive decline in total lung capacity (TLC) and vital capacity, along with impairment of diffusion capacity and subsequent development of (primarily hypoxic) respiratory failure along with respiratory muscle dysfunction.

Studies have supported the advantage of ultrasonography in the assessment of diaphragmatic mobility by two-dimensional (BD) or M-mode. Others reported the investigation methods, the criteria for normal and pathological diaphragmatic function, and the perspectives of development in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* patients presented to Ain Shams University Hospital outpatient clinic by ILD due to any cause

Exclusion Criteria:

* Pregnant females
* Patients with end stage organ failure e.g.: Renal failure, liver cell failure
* Patients with malignancy elsewhere.
* The patients who refuse to be entitled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presented to Ain Shams University Hospital's chest outpatient clinic by ILD due to any cause with age more than 18 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
diaphragm mobility assessment in different types of interstitial lung diseases | 1 year
  measurement of diaphragmatic excursion in cm in different types of interstitial lung diseases

SECONDARY OUTCOMES:
Correlation between diaphragmatic mobility and functional assessment in different ILD types | 1 year
  find the correlation between excursion measurements and spirometry indices, DLCO and CT fibrosis score

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
no IPD will be shared